CLINICAL TRIAL: NCT03424213
Title: Race-related Alternative Splicing: Novel Targets in Prostate Cancer
Acronym: PCaP splicing
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00091092
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — radical prostatectomy specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- white low aggressive: low aggressive = Gleason score < 7 and stage cT1-cT2 and PSA < 10 ng/ml
  Interventions: Other: No interventions - retrospective data collection
- white high aggressive: high aggressive = Gleason score ≥ 8 or PSA > 20 ng/ml or Gleason score = 7 and stage cT3-cT4
  Interventions: Other: No interventions - retrospective data collection
- white intermediate aggressive: intermediate aggressive = all other cases
  Interventions: Other: No interventions - retrospective data collection
- AA low aggressive: low aggressive = Gleason score < 7 and stage cT1-cT2 and PSA < 10 ng/ml
  Interventions: Other: No interventions - retrospective data collection
- AA high aggressive: high aggressive = Gleason score ≥ 8 or PSA > 20 ng/ml or Gleason score = 7 and stage cT3-cT4
  Interventions: Other: No interventions - retrospective data collection
- AA intermediate aggressive: intermediate aggressive = all other cases
  Interventions: Other: No interventions - retrospective data collection

INTERVENTIONS:
Other: No interventions - retrospective data collection — No new patients will be consented to this study. Only retrospective data will be collected on prostatectomy specimens and correlated with health data

SUMMARY:
Data from evaluating prostate cancer (PCa) biopsy tissue from AA and white patients has led to the discovery of alternative splicing as a novel molecular mechanism underlying more aggressive PCa in AA men. Coded archival radical prostatectomy tissue specimens and annotated clinical data, questionnaire data, and ancestral genotyping data will be obtained from the racially diverse and federally funded North Carolina-Louisiana PCa Project (NC-LA PCaP). We will use 33 tissue specimens from each of the following 6 groups (n=198 total): white low aggressive, white intermediate aggressive, white high aggressive, AA low aggressive, AA intermediate aggressive and AA high aggressive. The aforementioned tissues will first be screened for tumor content and Gleason grade by a genitourinary pathologist. To identify race-related splice variants, RNA will be isolated for targeted sequencing of prioritized race-related alternatively spliced genes using the NimbleGen SeqCap Target Enrichment, SeqCap RNA System to capture regions of interest and the Illumina HiSeq sequencing platform to sequence these regions at a depth and coverage sufficient to accurately call alternative splicing events.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of prostate cancer.
2. Self-reported race of AA or white.
3. Availability of five unstained slides per radical prostatectomy specimen and an associated Hematoxylin and Eosin stained slide for each radical prostatectomy specimen from NC-LA PCaP.
4. Classification of prostate cancer of low, intermediate or high aggressiveness, as defined by NC-LA PCaP.

Exclusion Criteria:

1. Obtained radical prostatectomy tissue is inadequate for RNA analysis and/or is not positive for adenocarcinoma of the prostate of low, intermediate or high aggressiveness.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes AA and white male patients having confirmed prostate cancer and enrolled in NC-LA PCaP, a population-based, case-only study of prostate cancer in AA and white men in NC and LA. Radical prostatectomy specimens will be selected from AA and white patients who have consented to NC-LA PCaP and have adequate tumor specimens of appropriate aggressiveness banked.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Frequency of candidate race-related splice variants in localized prostate cancer of varying degrees of aggressiveness | at the time of analysis

CONTACTS AND LOCATIONS:
Overall Officials: Steve Patierno, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No